CLINICAL TRIAL: NCT00326287
Title: A Randomized, Double-Blind, Multicenter Study of Ceftobiprole Medocaril Versus Placebo in the Treatment of Subjects Hospitalized With Community-Acquired Pneumonia
Brief Title: Ceftobiprole in the Treatment of Patients With Community-Acquired Pneumonia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR011407; 30982081-CAP-3001 (Other: Basilea Pharmaceutica International Ltd.)
Record Dates: First submitted 2006-05-12; First posted 2006-05-16 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-07

CONDITIONS: Pneumonia
Keywords: Community-Acquired Pneumonia; Cephalosporins; Methicillin-Resistant Staphylococcus Aureus
MeSH Terms: conditions — Pneumonia; Community-Acquired Pneumonia | interventions — ceftobiprole medocaril; Ceftriaxone; Linezolid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ceftobiprole medocaril (Experimental): Ceftobiprole medocaril 500mg q8h as 2h infusions, 7-14d
  Interventions: Drug: Ceftobiprole medocaril
- Ceftriaxone with or without Linezolid (Active Comparator): Ceftriaxone 2g qd as 0.5h infusions with or without Linezolid 600mg q12h as 1h infusions, 7-14d
  Interventions: Drug: Ceftriaxone with or without Linezolid

INTERVENTIONS:
Drug: Ceftobiprole medocaril
  Arms: Ceftobiprole medocaril
Drug: Ceftriaxone with or without Linezolid
  Arms: Ceftriaxone with or without Linezolid

SUMMARY:
The purpose of this study is to compare the clinical cure rate (ratio of clinically cured patients to the total number of patients) of ceftobiprole medocaril versus a comparator in the treatment of patients with community-acquired pneumonia.

DETAILED DESCRIPTION:
Ceftobiprole medocaril is a cephalosporin antibiotic with anti-MRSA (Methicillin-Resistant Staphylococcus Aureus) activity. Ceftobiprole medocaril is not yet approved for the treatment of community-acquired pneumonia. This is a randomized, double-blind, multicenter study of ceftobiprole medocaril plus placebo versus a comparator to assess the effectiveness and safety of ceftobiprole medocaril in patients with community-acquired pneumonia. The patients will be randomized to ceftobiprole medocaril plus placebo or a comparator. Patients who meet specified criteria may be switched to an alternative oral treatment. The primary endpoint is that the clinical cure rate among patients treated with ceftobiprole at the test of cure visit. The patients will receive either ceftobiprole medocaril plus placebo or a comparator.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from community-acquired pneumonia severe enough to require hospitalization
* Female patients must be postmenopausal for at least 1 year, surgically sterile, or practicing an effective method of birth control before entry and throughout the study

Exclusion Criteria:

* Patients with known or suspected hypersensitivity to any related antibiotic medications
* Treatment with any experimental drug within 30 days before enrollment
* Prior enrollment in this study or any study with ceftobiprole medocaril

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 638 (Actual)
Dates: Start 2006-06; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Clinical cure rate (ratio of the number of clinically cured patients to the total number of patients) at the test of cure visit that occurs 7 to 14 days after the last dose of study drug | 7 weeks

SECONDARY OUTCOMES:
Microbiological eradication rate (ratio of the number of patients with microbiological eradication to the total number of patients) | 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Huang H, Gao L, Engelhardt M, Saulay M, Hamed K. A post hoc analysis of two Phase III trials showing the efficacy and tolerability of ceftobiprole in East Asian patients. Future Microbiol. 2021 Jul;16:783-796. doi: 10.2217/fmb-2021-0121. Epub 2021 Jun 22. PMID 34155899
- [Derived] Welte T, Scheeren TW, Overcash JS, Saulay M, Engelhardt M, Hamed K. Efficacy and safety of ceftobiprole in patients aged 65 years or older: a post hoc analysis of three Phase III studies. Future Microbiol. 2021 May;16:543-555. doi: 10.2217/fmb-2021-0042. Epub 2021 May 7. PMID 33960817
- [Derived] Scheeren TWL, Welte T, Saulay M, Engelhardt M, Santerre-Henriksen A, Hamed K. Early improvement in severely ill patients with pneumonia treated with ceftobiprole: a retrospective analysis of two major trials. BMC Infect Dis. 2019 Feb 26;19(1):195. doi: 10.1186/s12879-019-3820-y. PMID 30808293
- [Derived] Nicholson SC, Welte T, File TM Jr, Strauss RS, Michiels B, Kaul P, Balis D, Arbit D, Amsler K, Noel GJ. A randomised, double-blind trial comparing ceftobiprole medocaril with ceftriaxone with or without linezolid for the treatment of patients with community-acquired pneumonia requiring hospitalisation. Int J Antimicrob Agents. 2012 Mar;39(3):240-6. doi: 10.1016/j.ijantimicag.2011.11.005. Epub 2012 Jan 9. PMID 22230331
- See also: Ceftobiprole in the Treatment of Patients with Community-Acquired Pneumonia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=731&filename=CR011407_CSR.pdf.pdf